CLINICAL TRIAL: NCT01346735
Title: Multi-center Observational Study to Evaluate Epidemiology and Resistance Patterns of Common ICU-Infections (MOSER)
Acronym: MOSER
Status: Completed | Type: Observational
Sponsor: Indian Society of Critical Care Medicine (Other)
Responsible Party: Principal Investigator, Dr. Ramesh Venkataraman, Dr, Indian Society of Critical Care Medicine
Other Study IDs: ISCCM1
Record Dates: First submitted 2011-05-02; First posted 2011-05-03 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Nosocomial Infections
Keywords: Ventilator associated pneumonia; Catheter related blood stream infection; Catheter associated urinary tract infection; ICU-related infections (VAP, CAUTI and CRBSI); India
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ICU infections: Infections acquired during the ICU stay
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Most literature on ICU infections and the resistant patterns comes from the western literature. This data may not truly reflect the incidence, epidemiology and resistance patterns in developing countries such as India. However, empiric antibiotic therapy is generally initiated using western guidelines. This can potentially lead to inadequate, inappropriate and ineffective empiric antibiotic therapy for ICU infections in the Indian setting. Hence in this multi-center observational study, we seek to:

1. To determine the incidence of ICU-related infections (VAP, CAUTI and CRBSI) in India
2. To explore the microbiology, resistance and treatment patterns of these infections

ELIGIBILITY:
Inclusion Criteria:

1. ICU stay >48 hours
2. One of the following infections (VAP, CAUTI or CRBSI)

Exclusion Criteria:

1. Index ICU stay < 48 hours
2. Re-admissions to the ICU within the same hospitalization
3. Age >18 years or <70 years
4. Known HIV serology positivity
5. Burns
6. Solid organ or Bone-marrow transplant
7. No ICU-acquired infections (specifically VAP, CAUTI and CRBSI)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 381 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indian Society of Critical Care Medicine, Mumbai, India